CLINICAL TRIAL: NCT03270566
Title: An Outcome Assessor-blinded Pilot Randomised Controlled Trial of an Ion-exchange Water Softener for the Prevention of Atopic Eczema in Neonates, With an Embedded Mechanistic Study
Brief Title: Softened Water for Eczema Prevention Pilot Trial
Acronym: SOFTER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); University of Nottingham (Other); University of Sheffield (Other); Imperial College London (Other); University of Amsterdam (Other); University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRAS 233005
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-08

CONDITIONS: Atopic Eczema
Keywords: Water hardness; Atopic eczema prevention; Skin barrier function; Skin microbiome
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Domestic ion-exchange water softener (Experimental): The intervention group will have a domestic ion-exchange water softener installed prior to birth.
  Interventions: Device: Domestic ion-exchange water softener
- Usual hard water supply (No Intervention): The control group will receive their usual domestic water supply.

INTERVENTIONS:
Device: Domestic ion-exchange water softener — Ion-exchange water softeners exchange calcium and magnesium, amongst other divalent cations, for monovalent sodium cations using a polystyrene resin. The sodium ions come from sodium chloride (common salt). The salt needs to be topped up every 3-4 weeks and sufficient quantities of block salt will be supplied to participants. The water softener used in this study does not require electricity and has two cylinders of resin which are used alternately. A control valve alternates the flow between the two cylinders and ensures a constant supply of regenerated resin. Ion-exchange water softeners typically reduce downstream water hardness to close to zero.
  Arms: Domestic ion-exchange water softener

SUMMARY:
An outcome assessor-blinded pilot randomised controlled trial of an ion-exchange water softener for the prevention of atopic eczema in neonates, with an embedded mechanistic study

DETAILED DESCRIPTION:
A 6-month parallel group assessor-blinded pilot randomised controlled trial of an ion-exchange water softener for the prevention of eczema in neonates, with an embedded mechanistic study.

The overall rationale is that by installing a domestic water softener around the time of birth, the infant will be exposed to softened water rather than hard water for bathing and that this will be less irritating to the skin than hard water and so associated with a lower risk of eczema development. The primary objective is to determine the feasibility of conducting a subsequent definitive RCT that will investigate whether installation of a domestic water softener around the time of birth can prevent eczema in high-risk babies. The secondary objective is to explore the likely mechanisms by which water softeners might prevent eczema.

ELIGIBILITY:
Inclusion Criteria:

* Participant (i.e. the neonate) must have a parent or sibling with a history of doctor-diagnosed atopy (i.e. at least one of: eczema, asthma, hayfever)
* Mother aged ≥18 years of age at enrolment
* Baby <36 weeks gestation at screening
* Informed consent from the mother on behalf of the participant
* Mother has the ability to understand English
* Live in a hard water area (>250 mg/L Calcium Carbonate)
* Consent of landlord for installation on water softener (if appropriate)
* Occupy a property appropriate for installation of a water softener

Exclusion Criteria:

* Preterm birth (defined as birth prior to 37 weeks gestation)
* Significant inflammatory skin disease at birth not including seborrheic dermatitis ("cradle cap")
* Sibling (including twin) previously randomised to this trial. If multiple birth, the first child will be randomised into the trial.
* The child is to be fostered/adopted
* Any immunodeficiency disorder or severe genetic skin disorder
* Child has any other serious health issue which, at parent or investigator discretion, would make it difficult for the family to take part in the trial.
* Planned stays away from home for a continuous period of more than 2 weeks or a total of 1 month out of the 6 month follow up period
* Water softening or filtration device already installed
* Concurrent enrolment in any other skin-related intervention study
* Other medical condition that in the opinion of the CI could interfere with the conduct of the trial

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible families screened who are willing and able to be randomised. | Before birth
  This is key to the determination of the likely success of a future, large-scale definitive randomised controlled trial (RCT).

SECONDARY OUTCOMES:
Proportion of pregnant women approached who agree to be screened | Before birth
Proportion of families eligible on screening that cannot have a water softener installed (e.g. due to landlord or local authority refusal, technical (plumbing) reasons) | Before birth
Proportion of families randomised that withdraw due to infant ineligibility | Baseline (birth)
Proportion of families in intervention arm who found the intervention acceptable | End of follow up (6 months of age)
Proportion of participants in control arm that become exposed to softened water | End of follow up (6 months of age)
  (e.g. by moving to a new home in a soft water area, or moving to a home with an active water softener installed, before the end of follow up)
Proportion of participants that have the water softening unit removed or disabled prior to end of follow up | End of follow up (6 months of age)
Proportion of participants with visible eczema status (yes/no) recorded | Baseline, 4 weeks, 3 and 6 months
  According to UK diagnostic criteria-based photographic protocol
Proportion of water samples with hardness >20 mg/L calcium carbonate | Between installation and end of follow up
  Would suggest failure of the water softening device
Proportion of participants that withdraw from the trial prior to end of follow up | From randomisation until end of follow up
Median number of nights spent away from the participant's main home during follow up | From birth until end of follow up (6 months of age)
Proportion of clinical outcome assessments that have remained blinded | at 4 weeks, 3 & 6 months
Proportion with patient-reported, doctor-diagnosed eczema | by 6 months of age
Proportion with visible eczema according to the UK diagnostic criteria-based photographic protocol | 4 weeks, 3 & 6 months
Severity of eczema (if present) using Eczema Area and Severity Index (EASI) | 4 weeks, 3 & 6 months
Patient-reported eczema symptoms (Patient-Orientated Eczema Measure - POEM) | Monthly from 4 weeks to 6 months of age
Time to onset of patient-reported doctor-diagnosed eczema | from birth to end of follow up (6 months of age)

OTHER OUTCOMES:
Transepidermal water loss (TEWL) | at birth, 4 weeks, 3 & 6 months oif age
Cutaneous cytokine profiles | at birth, 4 weeks, 3 & 6 months oif age
  e.g. interleukin-1 levels
Natural moisturising factor (NMF) levels | at birth, 4 weeks, 3 & 6 months oif age
Shannon Diversity Index and other skin and respiratory microbiota parameters | at birth, 4 weeks, 3 & 6 months oif age
Proportion with filaggrin null mutations | at birth, 4 weeks, 3 & 6 months oif age
Effect of filaggrin (FLG) gene mutation status on TEWL, cytokine levels, NMF levels and skin microbiota diversity | at birth, 4 weeks, 3 & 6 months oif age
Median domestic water hardness level (calcium carbonate concentration) | at birth, 4 weeks, 3 & 6 months oif age
Skin hydration | at birth, 4 weeks, 3 & 6 months oif age

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Flohr, PhD, FRCPCH, Principal Investigator — King's College London
Locations (1):
- St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD

REFERENCES:
- [Derived] Jabbar-Lopez ZK, Ezzamouri B, Briley A, Greenblatt D, Gurung N, Chalmers JR, Thomas KS, Frost T, Kezic S, Common JEA, Danby S, Cork MJ, Peacock JL, Flohr C. Randomized controlled pilot trial with ion-exchange water softeners to prevent eczema (SOFTER trial). Clin Exp Allergy. 2022 Mar;52(3):405-415. doi: 10.1111/cea.14071. Epub 2021 Dec 12. PMID 34854157
- [Derived] Laughter MR, Maymone MBC, Mashayekhi S, Arents BWM, Karimkhani C, Langan SM, Dellavalle RP, Flohr C. The global burden of atopic dermatitis: lessons from the Global Burden of Disease Study 1990-2017. Br J Dermatol. 2021 Feb;184(2):304-309. doi: 10.1111/bjd.19580. Epub 2020 Nov 29. PMID 33006135
- [Derived] Jabbar-Lopez ZK, Gurung N, Greenblatt D, Briley A, Chalmers JR, Thomas KS, Frost T, Kezic S, Common JEA, Kong HH, Segre JA, Danby S, Cork MJ, Peacock JL, Flohr C. Protocol for an outcome assessor-blinded pilot randomised controlled trial of an ion-exchange water softener for the prevention of atopic eczema in neonates, with an embedded mechanistic study: the Softened Water for Eczema Prevention (SOFTER) trial. BMJ Open. 2019 Aug 20;9(8):e027168. doi: 10.1136/bmjopen-2018-027168. PMID 31434765